CLINICAL TRIAL: NCT01074645
Title: Tenofovir Reduces Morbidity and Mortality in Patients With Spontaneous Reactivation of Hepatitis B Presenting as Acute-on-chronic Liver Failure (ACLF): A Randomized Placebo Controlled Trial
Brief Title: Randomized Controlled Trial of Tenofovir in Patients of Reactivation of Hepatitis B Presenting as Acute on Chronic Liver Failure
Acronym: ACLF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Shiv K Sarin, G.B. Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hitendra garg
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2009-10

CONDITIONS: Acute on Chronic Liver Failure; Hepatitis B
Keywords: Acute-on -chronic liver failure; Reactivation of hepatitis B; Spontaneous reactivation of chronic hepatitis B presenting as to acute-on-chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (No Intervention): Placebo was the multivitamin capsule which was similar in appearance as of Tenofovir disoproxil fumarate and was given once a day till 3 month.
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)
- Tenofovir disoproxil fumarate (TDF) (Active Comparator): Tenofovir disoproxil fumarate (TDF) is a potent, rapidly acting, oral acyclic nucleotide analogue, reverse transcriptase inhibitor that has been shown to be highly effective in suppressing hepatitis B virus replication. Tenofovir has also shown excellent activity against HBV in both LAM- naïve and LAM-resistant patients. Its efficacy has not been evaluated in patients of reactivation of hepatitis B who present as ACLF
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (TDF) — Tenofovir 300mg/day for 3 month

SUMMARY:
Background: Reactivation of hepatitis B is a well-characterized syndrome marked by the abrupt reappearance or rise of hepatitis B virus (HBV) DNA in the serum of a patient with previously inactive or resolved HBV infection. Reactivation can be spontaneous, but is most commonly triggered by cancer chemotherapy, immune suppression, or alteration in immune function. Spontaneous acute exacerbation of chronic hepatitis B infection is seen with a cumulative probability of 15±37% after 4 years of follow-up.2 Significant number of patients of spontaneous acute exacerbation of chronic hepatitis B may present with very high ALT levels, jaundice and liver failure.3 This condition should be defined as acute-on-chronic liver failure (ACLF) according to a recent Asia-Pacific consensus recommendation.

The short term prognosis of patients of spontaneous acute exacerbation of chronic hepatitis B leading to ACLF like presentation is extremely poor, with a mortality of 30-70% in different series.8,9,10 Liver transplantation has been the only definitive therapy available to salvage this group of patients. However ,this is not readily available and affordable. Another therapeutic option is antiviral therapy but has limited data. The efficacy of lamivudine was evaluated and compared by historical control but was not found to be beneficial.8,9,10 However ,a study from Taiwan showed a survival benefit in a subgroup of patients who were on lamivudine and had baseline bilirubin below 342 mmol/L (20 mg/dL).11 Tenofovir disoproxil fumarate (TDF) is a potent, rapidly acting, oral acyclic nucleotide analogue, reverse transcriptase inhibitor that has been shown to be highly effective in suppressing hepatitis B virus replication.12 Tenofovir has also shown excellent activity against HBV in both LAM- naïve and LAM-resistant patients.13,14. Its efficacy has not been evaluated in patients of reactivation of hepatitis B who present as ACLF Hypothesis: The investigators hypothesis that Tenofovir reduces the morbidity and mortality in patients with Spontaneous reactivation of hepatitis B by reducing HBV DNA.

ELIGIBILITY:
Inclusion Criteria:

* Reactivation of chronic hepatitis B characterized by rise in ALT level >5 times upper limit of normal along with HBV DNA level >105 copies/ml (~1.8x104 IU/ml) presenting as ACLF
* Acute hepatic insult
* Jaundice (bilirubin ≥5 mg/dL) and coagulopathy (INR>1.5)
* Complicated within 4 weeks by ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease.

Exclusion Criteria:

* Superinfection with other viruses (Hepatitis E, A, D and C)
* Coexistent hepatocellular carcinoma (HCC)
* Portal vein thrombosis
* Coexistent renal impairment
* Pregnancy
* Co-infection with HIV infection or Patients received previous course of any antiviral
* Immunomodulator or cytotoxic/immunosuppressive therapy for chronic hepatitis or other illness within at least the preceding 12 month.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reduction in HBV DNA levels, survival | 3 Month

SECONDARY OUTCOMES:
Improvement in CTP, MELD scores | 3 Month

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD,DM, Principal Investigator — G.B. Pant Hospital, New Delhi, India
Locations (1):
- Department of Gastroenterology, GB Pant Hospital,, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Garg H, Sarin SK, Kumar M, Garg V, Sharma BC, Kumar A. Tenofovir improves the outcome in patients with spontaneous reactivation of hepatitis B presenting as acute-on-chronic liver failure. Hepatology. 2011 Mar;53(3):774-80. doi: 10.1002/hep.24109. Epub 2011 Feb 3. PMID 21294143